CLINICAL TRIAL: NCT02196636
Title: A Single-center, Randomised, Double-blind, Adaptative, Parallel Study to Investigate the Safety, Tolerability, Pharmacokinetics (Including the Effect of Food), and Pharmacodynamics or RO6806127 in Healthy Male Subjects
Brief Title: A Phase 1 Study of RO6806127 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BP29276; 2014-001019-38 (EudraCT Number)
Record Dates: First submitted 2014-07-16; First posted 2014-07-22 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Part 1: Single Ascending Dose (SAD) (Experimental): Adaptive model per protocol
  Interventions: Drug: Placebo; Drug: RO6806127
- Part 2: Food Effect (FE) (Experimental): Fasted versus Fed
  Interventions: Drug: Placebo; Drug: RO6806127

INTERVENTIONS:
Drug: Placebo — Matching placebo, administered orally with approximately 240 mL of buffer
Drug: RO6806127 — Administered orally with approximately 240 mL of buffer

SUMMARY:
This two-part study will assess the safety and tolerability of single ascending oral doses of RO6806127 in a group of healthy male participants and investigate the effect of high fat and high caloric food on the relative bioavailability of a single oral dose of RO6806127 in a separate group of healthy male participants. The relationship between drug exposure and tolerability will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants aged 18 to 45 years, inclusive
* A BMI between 18 to 30 kg/m2, inclusive
* Agreement to use highly effective contraception

Exclusion Criteria:

* Clinically significant abnormalities in laboratory test results
* History of any clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardio-vascular, endocrinological, hematological or allergic disease, metabolic disorder, cancer or cirrhosis
* Significant disorders of the central nervous system, including psychiatric disorders, behavioral disturbances, cerebrovascular events, depression, bipolar disorder, migraine, Parkinson, anxiety, any personal or familial history of seizures, epilepsy or other convulsive condition, previous significant head trauma, or other factors predisposing to seizures
* Use of any prohibited medications and food before study start and during the study
* Dietary restrictions that would prohibit the consumption of standardized meals

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to Day 21

SECONDARY OUTCOMES:
Phamacokinetic profile of single-dose oral RO6806127 and its metabolites as appropriate, as assessed by concentrations over time in plasma and urine | Up to Day 21
RO6806127 metabolite concentrations in selected plasma and urine samples | Up to Day 21
Relative bioavailability (food effect): Area under the concentration-time curves [AUC] | Up to Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Marlton, New Jersey, United States